CLINICAL TRIAL: NCT03005548
Title: Cortical Modulation of Acute Post-thoracotomy Pain With Transcranial Direct Current Stimulation
Acronym: CMAPTPtDCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Military Medical Academy, Belgrade, Serbia (Other)
Responsible Party: Principal Investigator, Dusica Stamenkovic, Associate Professor, MD, PhD, Anesthesiologist, Military Medical Academy, Belgrade, Serbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MF-VMA// 07.12.2015.
Record Dates: First submitted 2016-12-24; First posted 2016-12-29 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative
Keywords: Transcranial Direct Current Stimulation; Pain Postoperative; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Transcranial Direct Current Stimulation; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Experimental): Experimental: Transcranial direct current stimulation (tDCS). Patients assigned to the active treatment group (n=31) will receive IV morphine followed by IV morphine PCA (IV morphine bolus 1 mg, lockout time 10 mins.), preceded by tDCS (20 minutes of 2 milliamperes (mA) anodal tDCS over the ipsilateral cortex for 5days/week).
  Interventions: Device: Transcranial direct current stimulation; Drug: Morphine
- Sham tDCS (Sham Comparator): Sham Control Group: Patients assigned to the control group (n=31) will receive IV morphine followed by IV morphine PCA (IV morphine bolus 1 mg, lockout time 10 mins.), preceded by sham tDCS stimulation (30 sec over the ipsilateral cortex, 5 days/week).
  Interventions: Drug: Morphine

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation. All eligible patients will be treated with patient-controlled IV morphine analgesia by PCA (PCA pump (CADD-Legacy PCA Pump, Deltec, Inc.) IV morphine bolus 1 mg, lockout time 10 mins.).
  Device: wireless tDCS (StarStim, NeuroElectrics) non-invasive brain stimulation with a pair of electrodes with saline-soaked pads for delivery of direct current at intensity 2 mA for 20 mins.
  Other Names: tDCS
  Arms: Active tDCS
Drug: Morphine — In Sham comparator group All eligible patients will be treated with patient-controlled IV morphine analgesia (PCA) (PCA pump (CADD-Legacy PCA Pump (Deltec, Inc.) morphine IV bolus 1 mg, lockout time 10 mins).
  Device: wireless tDCS (StarStim, NeuroElectrics) non-invasive brain stimulation with a pair of electrodes with saline-soaked pads for delivery of direct current at intensity 2 mA for 30s at the beginning.

SUMMARY:
The primary objective of this single center, prospective, randomized, double blind clinical trial is to evaluate the effectiveness of anodal transcranial direct current stimulation (tDCS) combined with patient controlled analgesia (PCA) morphine, on intravenous morphine use for postoperative analgesia after thoracotomy. The intervention group will receive treatment with anodal tDCS, whereas the control group will receive sham stimulation.

DETAILED DESCRIPTION:
tDCS has been used for treatment of chronic pain states, but experience with the use of tDCS for treatment of acute postoperative pain is limited. tDCS has been used for postoperative analgesia after lumbar spine surgery, total knee arthroplasty and for post-procedural pain after endoscopic retrograde cholangiopancreatography.

This study investigates the effects of tDCS vs. sham stimulation combined with IV morphine PCA on postoperative morphine consumption for analgesia after thoracotomy for lung cancer.

Patients with malignant lung disease requiring thoracotomy will be randomly assigned to active stimulation or sham stimulation in a double-blind, sham-controlled, parallel design clinical trial. Each group will receive IV morphine PCA and tDCS vs. IV morphine PCA and sham stimulation daily, starting with arrival in the post-anesthesia care unit on the day of surgery and continuing for the first four postoperative days. Anodal tDCS with direct current at intensity 2 mA will be delivered for 20 minutes on five consecutive days, whereas sham stimulation will last for 30 seconds.

Morphine consumption, the number of analgesia demands, and pain intensity at rest, during movement and with cough will be recorded at predetermined time intervals as follows: After surgery, when VAS pain score at rest falls below 30 mm, tDCS will be applied. VAS pain will be measured immediately before the intervention (T0) and immediately after the intervention (T1), and then regularly every one hour for the four hours (Т2-Т5), and then every six hours (Т6-Т9) for five days.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide written informed consent,
* Subject is 18-80 years old,
* Subject needs thoracotomy for confirmed malignant lung disease,
* Subject is extubated in the operating room

Exclusion Criteria:

* Subject is pregnant
* Subject is in treatment for psychiatric disease
* Subject is in treatment for neurological disease
* Subject is in treatment for chronic pain
* Subject has history of current or past alcohol or Street Drug abuse
* Subject has received chemotherapy
* Subject has history of previous thoracic or cardiac surgery
* Subject is allergic to medications that will be used in the study
* Subject has pacemaker or automatic implantable cardioverter/defibrillator
* Subject has implants or any other devices in the head, the spinal cord or peripheral nerves
* Subject has confirmed brain lesion, including tumor or metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Amount of morphine used for treatment of pain after thoracotomy in a group of patients receiving tDCS combined with intravenous morphine PCA compared with a group of patients receiving sham stimulation combined with intravenous morphine PCA. | Five days
  Daily during five postoperative days

SECONDARY OUTCOMES:
Pain scores measured using visual analogue scale (VAS) at rest, during movement and during cough in patients receiving tDCS combined and IV morphine PCA compared with patients receiving sham stimulation and IV morphine PCA. | Five days
  After surgery, when VAS pain score at rest falls below 30 mm, tDCS will be applied. VAS pain will be measured immediately before the intervention (T0) and immediately after the intervention (T1), and then regularly every one hour for the four hours (Т2-Т5), and then every six hours (Т6-Т9) for five days.

CONTACTS AND LOCATIONS:
Overall Officials: Tihomir V Ilic, MD, PhD, Study Chair — Military Medical Academy, Bulgaria; Dusica M Stamenkovic, MD, PhD, Principal Investigator — Military Medical Academy, Bulgaria
Locations (1):
- Military Medical Academy, Department of Anesthesiology, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dubois PE, Ossemann M, de Fays K, De Bue P, Gourdin M, Jamart J, Vandermeeren Y. Postoperative analgesic effect of transcranial direct current stimulation in lumbar spine surgery: a randomized control trial. Clin J Pain. 2013 Aug;29(8):696-701. doi: 10.1097/AJP.0b013e31826fb302. PMID 23719070
- [Result] Borckardt JJ, Reeves ST, Robinson SM, May JT, Epperson TI, Gunselman RJ, Schutte HD, Demos HA, Madan A, Fredrich S, George MS. Transcranial direct current stimulation (tDCS) reduces postsurgical opioid consumption in total knee arthroplasty (TKA). Clin J Pain. 2013 Nov;29(11):925-8. doi: 10.1097/AJP.0b013e31827e32be. PMID 23370085
- [Result] Borckardt JJ, Romagnuolo J, Reeves ST, Madan A, Frohman H, Beam W, George MS. Feasibility, safety, and effectiveness of transcranial direct current stimulation for decreasing post-ERCP pain: a randomized, sham-controlled, pilot study. Gastrointest Endosc. 2011 Jun;73(6):1158-64. doi: 10.1016/j.gie.2011.01.050. Epub 2011 Apr 5. PMID 21470608
- [Derived] Stamenkovic DM, Mladenovic K, Rancic N, Cvijanovic V, Maric N, Neskovic V, Zeba S, Karanikolas M, Ilic TV. Effect of Transcranial Direct Current Stimulation Combined With Patient-Controlled Intravenous Morphine Analgesia on Analgesic Use and Post-Thoracotomy Pain. A Prospective, Randomized, Double-Blind, Sham-Controlled, Proof-of-Concept Clinical Trial. Front Pharmacol. 2020 Feb 25;11:125. doi: 10.3389/fphar.2020.00125. eCollection 2020. PMID 32161547